CLINICAL TRIAL: NCT05069623
Title: A Phase 1/2, Open Label, Dose Escalation Study to Determine Safety and Immunogenicity of Two (Prophylactic) COVID 19 DNA Vaccine Candidates (VB10.2129 [C1], a RBD Candidate and VB10.2210 [C2], a T Cell Candidate), in Healthy Adult Volunteers
Brief Title: A Phase 1/2 Study to Determine Safety and Immunogenicity of Two COVID 19 Vaccines VB10.2129 (RBD Candidate) and VB10.2210 (T Cell Candidate) Previously Vaccinated in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nykode Therapeutics ASA (Industry)
Collaborators: Vaccibody AS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VB-D-01
Record Dates: First submitted 2021-10-04; First posted 2021-10-06 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; Infection Viral; Infections
Keywords: COVID-19; Coronavirus; DNA vaccine; Vaccine
MeSH Terms: conditions — COVID-19; Virus Diseases; Infections; Coronavirus Infections | interventions — VB10.COV-2 vaccine

STUDY DESIGN:
Intervention Model Description: Two vaccine candidates are investigated in parallell.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VB10.2129 Part 1 Dose escalaton (Experimental): 0.3 mg, 1 mg or 3 mg will be administered by two IM injections 21 days apart.
  Interventions: Biological: VB10.2129
- VB10.2210 Part 1 Dose escalation (Experimental): 0.3 mg, 1 mg or 3 mg will be administered by two IM injections 21 days apart.
  Interventions: Biological: VB10.2210
- VB10.2129 Part 2 Dose expansion (Experimental): The seleceted dose from Part 1 will be administered IM in a two-dose schedule.
  Interventions: Biological: VB10.2129
- VB10.2210 Part 2 Dose expansion (Experimental): The seleceted dose from Part 1 will be administed IM in a two-dose schedule.
  Interventions: Biological: VB10.2210

INTERVENTIONS:
Biological: VB10.2129 — 0.3 mg, 1 mg or 3 mg on Day 0 and Day 21 or 3 mg on Day 0
  Arms: VB10.2129 Part 1 Dose escalaton; VB10.2129 Part 2 Dose expansion
Biological: VB10.2210 — 3 doses (dose to be determined) on Day 0 and Day 21 or highest dose (TBD) on Day 0
  Arms: VB10.2210 Part 1 Dose escalation; VB10.2210 Part 2 Dose expansion

SUMMARY:
An open label, dose escalation, and dose expansion study to evaluate the safety, reactogenicity and immunogenicity of two SARS-CoV-2 DNA plasmid vaccine candidates, VB10.2129 (C1) and VB10.2210 (C2). tThree dose levels will be tested. IM administrations 21 days apart. Part 1 is a dose escalation phase and Part 2 is a dose expansion phase. In Part 2 a selected dose will be tested further in additional healty volunteers.

DETAILED DESCRIPTION:
This is an open label, dose escalation, and dose expansion study designed to evaluate the safety, reactogenicity and immunogenicity of two SARS-CoV-2 or COVID-19 DNA plasmid vaccine candidates, VB10.2129 (C1) and VB10.2210 (C2).

Part 1 is a dose escalation phase and Part 2 is a dose expansion phase and both vaccine candidates, ie, VB10.2129 (C1) and VB10.2210 (C2) will be tested.

Part 1 consist of two arms: one arm with each vaccine candidate and each arm investigating three escalating dose levels.

10 subjects previously vaccinated with an mRNA vaccine will be enrolled at each dose level. Each subject will receive two vaccinations 21 days apart (Day 0 and Day 21).

In Part 2 is a dose expansion phase with one arm for each candidate; VB10.2129 and VB10.2210, in previously vaccinated healthy subjects only. The dose to be investigated will be selected based on safety and inital immune response data from Part 1. All subjects will be folowed for up to 1 year after the first vaccination.

ELIGIBILITY:
Main inclusion criteria:

* Give informed consent by signing the Informed Consent Form (ICF)

SARS CoV 2 vaccination status for Part 1:

1. VB10.2129 (C1): have received 2 or 3 doses of an approved mRNA SARS CoV 2 vaccine, minimum 4.5 months (20 weeks) prior to Visit 1.
2. VB10.2210 (C2): have received 2 doses (primary vaccination) or 3 (primary and boost) doses of an approved mRNA SARS CoV 2 vaccine, minimum 8 weeks prior to Visit 1.

SARS CoV 2 vaccination status for Part 2:

VB10.2129 (C1) and VB10.2210 (C2) Vaccination status prior to Visit 1 will be decided based on data from Part 1.

* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions (eg, local law and regulations [county specific lock down rules] regarding COVID-19), and other requirements of the study.
* Healthy, in the clinical judgement of the Investigator, based on medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs (systolic/diastolic blood pressure, pulse rate, body temperature, respiratory rate), and clinical laboratory tests (blood chemistry, haematology, and urine chemistry) at Visit 0 (Screening).
* Women of childbearing potential (WOCBP) must have a negative pregnancy test and must agree to practice a highly effective form
* Agree not to be vaccinated with any other vaccine during the study until 28 days after receiving the last study vaccination
* Negative rtPCR-test for SARS-CoV-2

Main exclusion criteria:

* Have had any acute illness with or without fever, within 72 hours prior to the first vaccination
* Symptoms of upper respiratory infection, fever, persistent cough, shortness of breath, runny nose and breathing difficulties
* Breastfeeding or who plan to breastfeed during the study
* Have a known allergy, hypersensitivity, or intolerance to aminoglycosides
* Had any clinically significant or chronic medical condition or any major surgery within the past 5 years which
* Have any surgery planned during the study
* Had any chronic use of any systemic medications, including immunosuppressant's, oral corticosteroids or other immune-modifying drugs, within the 12 months prior to Screening
* Received any vaccination within the 28 days prior to Screening
* Received any prescription medicines (except hormonal contraception for WOCBP) within 14 days prior to Visit 0 (Screening) or over the counter medicines (except paracetamol and acetaminophen at a dose of (≤2 grams/day)) within 48 hours of Visit 0.
* Have a known history or a positive test of HIV 1 or 2, Hep B, or Hep C
* Have a positive rtPCR test for SARS-CoV-2 within 2 days of Screening
* Documented history of previous infection with SARS-CoV-2 and/or who have the presence of serum Ab indicative of a previous SARS-CoV-2 infection
* Have a history of hypersensitivity or have had a serious reaction to a previous vaccination
* Have any abnormality or permanent body art (eg, tattoo) that, would obstruct the ability to observe local reactions at the injection site.
* Have a condition known to put them at high risk for severe COVID-19, including those with any of the following risk factors: Hypertension, diabetes mellitus, chronic pulmonary disease, asthma, chronic liver disease, known stage 3 or worse chronic kidney disease
* Anticipating the need for immunosuppressive treatment within the next 6 months.

Other inclusion or exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence and frequency of local and systemic solicited adverse events (AEs) | Day 0 to Day 7 days after each vaccination
  As self reported in eDiary
Incidence and frequency of local and systemic unsolicited AEs | Day 0 to Day 49
  As elicited by investigator
Incidence and frequency of serious AEs (SAEs) | Day 0 to 1 year
  As elicited by investigator

SECONDARY OUTCOMES:
Humoral responses against SARS-CoV-2 | Day 0 (before Dose 1) up to 1 year
  Number participants with increase in Ab titre and neutralizing Ab responses after first and second vaccine and long term responses (VB10.2129)
Cellular responses (T-cell responses) to SARS-CoV-2 RBD epitopes by ELISpot | Day 0 (before Dose 1) up to 1 year
  Number of participants with change from baseline in Antigen-Specific T-cell cytokine production and long term T-cell responses

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Klinisk Forskningspost, Bergen
  - Oslo University Hospital Ullevål Sykehus, Dept. Infection Diseases, Oslo

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries and all collected IPD will be stripped of identifiers and may be made available upon request.
Supporting Information: ICF
Time Frame: Anonymous IPD may be shared following or during the publication of summary data. Archival data may be accessed for up to 25 years following the end of the study.
Access Criteria: Those who request the anonymous IPD must provide a plan of study explaining how the data will be used. Requests may be sent to the Central Contact Person. Requests will be reviewed based on the potential for the planned use of the IPD for advancing scientific knowledge and theory.